CLINICAL TRIAL: NCT07258368
Title: Comparative Effect of Gong Mobilization and Spencer Technique in the Management of Frozen Shoulder Among Diabetic Patients
Brief Title: Gong Mobilization Versus Spencer Technique for Diabetic Frozen Shoulder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/ Afshan Batool 02212
Record Dates: First submitted 2025-09-25; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Frozen Shoulder
Keywords: Diabetic; Spencer technique; Pain
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spencer Technique + Conventional Treatment (Experimental): The Spencer Technique is an osteopathic shoulder mobilization performed with the patient lying on the unaffected side and the therapist stabilizing the scapula while moving the humerus. It consists of a sequence of seven articulatory steps: shoulder extension, flexion, circumduction with compression, circumduction with traction, abduction with internal rotation, internal rotation (hand behind back), and abduction with external rotation. Each movement is performed rhythmically at the end range to stretch the joint capsule, improve mobility, and reduce pain (Frequency: Over the course of 3 days, the exercise was repeated 3 times per session). Conventional PT: Hot pack = 15 mins, Home Plan: Pendulum Stretch, Cross-Body Arm Reach, Towel Stretch, Finger Walk (Wall Climb), External Rotation Stretch, Shoulder Blade Squeeze, Overhead Shoulder Stretch.
  Interventions: Other: Spencer Technique + Conventional Treatment
- Gong Mobilization + Conventional Treatment (Experimental): The shoulder joint was turned upward as the patient was positioned in a side-lying posture. The patient had a 90-degree abduction of the shoulder to keep the humerus upright, and the elbow was 90 degrees flexed. Now the therapist held one hand of the patient to apply pressure to the humeral head from anterior to posterior while maintaining the position of the elbow at 90 degrees. The therapist then raised their own body while softly pushing on the shoulder joint's articular capsule. To retain the humerus' vertical axis, they achieved this while keeping shoulder abduction and elbow flexion at 90 degrees. The procedure was finished in about two to three minutes, and the articular capsule was gently squeezed for 10-15 seconds, and then relaxed for five seconds. After slightly stretching the capsule, the therapist applied gentle pressure with one hand on the shoulder joint from anterior to posterior. Maitland grades 3,4 then performed and then grade 4 approach for stretching for secs.
  Interventions: Other: Gong Mobilization + Conventional Treatment

INTERVENTIONS:
Other: Spencer Technique + Conventional Treatment — The Spencer Technique is an osteopathic shoulder mobilization performed with the patient lying on the unaffected side and the therapist stabilizing the scapula while moving the humerus. It consists of a sequence of seven articulatory steps: shoulder extension, flexion, circumduction with compression, circumduction with traction, abduction with internal rotation, internal rotation (hand behind back), and abduction with external rotation. Each movement is performed rhythmically at the end range to stretch the joint capsule, improve mobility, and reduce pain (Frequency: Over the course of 3 days, the exercise was repeated 3 times per session). Conventional PT: Hot pack = 15 mins, Home Plan: Pendulum Stretch, Cross-Body Arm Reach, Towel Stretch, Finger Walk (Wall Climb), External Rotation Stretch, Shoulder Blade Squeeze, Overhead Shoulder Stretch.
  Arms: Spencer Technique + Conventional Treatment
Other: Gong Mobilization + Conventional Treatment — The shoulder joint was turned upward as the patient was positioned in a side-lying posture. The patient had a 90-degree abduction of the shoulder to keep the humerus upright, and the elbow was 90 degrees flexed. Now the therapist held one hand of the patient to apply pressure to the humeral head from anterior to posterior while maintaining the position of the elbow at 90 degrees. The therapist then raised their own body while softly pushing on the shoulder joint's articular capsule. To retain the humerus' vertical axis, they achieved this while keeping shoulder abduction and elbow flexion at 90 degrees. The procedure was finished in about two to three minutes, and the articular capsule was gently squeezed for 10-15 seconds, and then relaxed for five seconds. After slightly stretching the capsule, the therapist applied gentle pressure with one hand on the shoulder joint from anterior to posterior. Maitland grades 3,4 then performed and then grade 4 approach for stretching for secs.
  Arms: Gong Mobilization + Conventional Treatment

SUMMARY:
The aim of this randomized controlled trial is to find the comparative effect of spencer technique and gong mobilization on pain, range of motion and functional disability among diabetic frozen shoulder patients.

DETAILED DESCRIPTION:
Frozen shoulder, also known as adhesive capsulitis, is a common musculoskeletal condition characterized by progressive pain, stiffness, and significant restriction of both active and passive range of motion in the shoulder joint. The condition typically progresses through three stages: the painful or freezing stage, marked by increasing pain and stiffness; the frozen or adhesive stage, where pain may subside but stiffness persists; and the thawing stage, during which mobility gradually improves. Risk factors include age, gender (more common in women), trauma, prolonged immobilization, and systemic conditions such as diabetes mellitus. Studies suggest Gong mobilization may offer superior ROM gains, while the Spencer technique provides significant long-term benefits, especially when combined with conventional therapy. Treatment effectiveness can vary, indicating a need for approaches tailored to individual patient factors and condition stage. This is particularly relevant for diabetic patients, who often experience slower, more complex recoveries.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HbA1c ≥6.5% will be included.
* Patients diagnosed with frozen shoulder stage II, will be included.

Exclusion Criteria:

* Receiving other clinical trials that could interfere with the outcomes of this study.
* Subject with recent history of surgery on affected shoulder
* Subject with history of any trauma/fracture around shoulder complex
* Subject with rotator cuff lesion and tendon calcification.
* Patients contraindicated to joint mobilization

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | 3 weeks
  It is a self-reported questionnaire designed to measure pain and functional disability in individuals with shoulder conditions, such as frozen shoulder or rotator cuff injuries. It consists of two subscales: pain and disability, providing a comprehensive assessment of shoulder function.
Numeric Pain Rating Scale | 3 weeks
  The NPRS is a segmented numeric version of the visual analog scale which is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Goniometer for range of motion | 3 weeks
  A goniometer is a standard clinical tool for objectively measuring joint range of motion (ROM). It demonstrates high validity, correlating strongly (r > 0.90) with advanced motion analysis systems. Its reliability is also excellent, with high intra-rater (ICC > 0.90) and inter-rater (ICC 0.85-0.99) scores. This makes it a dependable instrument for both assessing patients and guiding treatment in rehabilitation and research.

CONTACTS AND LOCATIONS:
Overall Officials: Maria khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- HBS General Hospital, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No